CLINICAL TRIAL: NCT04651296
Title: Efficacy of Mind-Body Approaches for the Treatment of Chronic Pain With Psychological Comorbidity
Brief Title: Compassion Meditation vs. Health Education for Veterans
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBC-010-20S; CX002041-01A2 (Other Grant/Funding Number: VA CSRD)
Record Dates: First submitted 2020-11-24; First posted 2020-12-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Stress Disorders, Posttraumatic; Depression
Keywords: meditation
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Intervention Model Description: Experimental condition: manualized compassion meditation protocol, a 10-session group-based meditation training class led by a trained instructor Control condition: manualized health education protocol, a 10-session group-based health education and discussion led by a trained instructor
Who Masked: Outcomes Assessor
Masking Description: The outcome evaluator is blind to experimental condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- compassion meditation (Experimental): 10 week, group-based manualized compassion meditation training
  Interventions: Behavioral: compassion meditation
- health education (Active Comparator): 10 week, group-based manualized health education protocol
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: compassion meditation — manualized compassion meditation training
  Other Names: cognitively-based compassion meditation for chronic pain with psychological comorbidity
  Arms: compassion meditation
Behavioral: health education — manualized health education group
  Other Names: health education while living with pain
  Arms: health education

SUMMARY:
Chronic pain (CP) is a major health problem for military Veterans, and CP is often associated with comorbid mental health problems, including posttraumatic stress disorder (PTSD) and depression. CP with psychological comorbidity is associated with increased healthcare costs, medication use, risk of suicide and rates of disability and reduced quality of life. Current empirically supported treatments do not always lead to substantial improvements (up to 50% of patients drop out or are do not respond to treatment). This project was designed to evaluate the efficacy of a novel intervention for addressing these challenges. Compassion meditation (CM), a meditative practice that focuses on the wish to remove suffering, is a contemplative practice that has promise for the amelioration of physical and mental health problems as well as promoting positive affect and improving quality of life. This study will evaluate the efficacy of Cognitively-Based Compassion Training for Chronic Pain with Psychological Comorbidity (CBCT-CP+) compared to Health Education while Living with Pain (H.E.L.P.) control condition, in a sample of among Veterans with CP conditions and psychological comorbidity.

DETAILED DESCRIPTION:
Chronic pain (CP), defined as persistent (>6 months), non-malignant, musculoskeletal or generalized pain, is a prevalent and costly public health problem. CP is highly prevalent among Veterans; 30-40% of Veterans have moderate to severe CP. CP has a significant negative impact on mental health and quality of life. CP is associated with declines in physical and social functioning, decreased activity levels, anxiety, negative mood, and depression. Approximately 1.6 million Veterans Health Administration (VHA) enrolled Veterans have CP and psychological distress associated with mental health comorbidities, including posttraumatic stress disorder (PTSD; ~50%), depression (~25%), and anxiety disorder(s) (~25%). Despite this urgent clinical need and extraordinary economic and societal costs, there are currently no evidence-based psychosocial interventions that simultaneously target comorbid mental health symptoms and CP interference in Veterans.

The Veterans Health Administration and National Center for Complementary and Integrative Health have similarly prioritized the use of complementary and integrative health approaches for the treatment of complex physical and mental health conditions. Currently, forty percent of Veterans with CP report using these approaches, and 70% of non-users would use these approaches if they were offered at the VA.

Compassion meditation (CM), a meditative practice that focuses on the wish to remove suffering, is a contemplative practice that has promise for the amelioration of physical and mental health problems as well as promoting positive affect and improving quality of life. CM has been shown to decrease anxiety and depressive symptoms in clinical populations, and is associated with reductions in pain severity, pain disability, pain catastrophizing, psychological distress, pain-related anxiety and depression, and pain-related anger in civilians with CP. CBCT (Cognitively-Based Compassion Training), a manualized CM protocol, is associated with reduced stress-related immune responses, improved negative affect, and reduced suicidality and depression in civilians. CBCT has also been shown to increase social connectedness and positive affect, and reduce depressive and PTSD symptoms in Veterans.

With this randomized controlled trial (RCT), the investigators will evaluate the efficacy of Cognitively-Based Compassion Training for Chronic Pain with Psychological Comorbidity (CBCT-CP+). The trial will compare CBCT-CP+ to Health Education while Living with Pain (H.E.L.P.) control condition, in a sample of 126 Veterans with CP conditions and psychological comorbidities. The rationale for the proposed study of compassion meditation for CP with psychological comorbidity is motivated by (1) a pressing clinical need, (2) a clear theoretical model, and (3) initial evidence of its safety, feasibility and potential positive clinical effect for improving psychiatric conditions among Veterans.

Findings from this study could inform clinical practice and policy by investigating whether a compassion-based intervention targeting both CP and psychological comorbidities will improve treatment outcomes for Veterans. Further, results of the trial will lay the groundwork for multi-site studies that would attempt to determine efficacy of CBCT-CP+ across VA clinics and formally investigate putative mechanisms of treatment effects. This work could ultimately lead to better care for Veterans, greater patient and therapist satisfaction, and lower healthcare and societal costs.

ELIGIBILITY:
Inclusion Criteria:

Criteria for inclusion include

* Veteran status
* age 18 or greater
* able to consent
* pain most days (> 3 days/week) for at least 6 months
* probable diagnosis of depression and/or PTSD

Exclusion Criteria:

* serious suicidality or homicidality that has required urgent or emergent evaluation or treatment within the past three months or a suicide attempt within the past year
* a known, untreated substance abuse or dependence problem (inclusion is possible if there is evidence that the individual has been afforded and is complying with treatment for the substance problem)
* untreated/unstable serious mental disorders, such as psychotic disorders or bipolar disorder, or serious dissociative symptoms
* cognitive impairment that would interfere with treatment, and
* concurrent enrollment in any other treatment specifically targeting chronic pain, anxiety, depression, or PTSD symptoms or social functioning (e.g., couples therapy) or any meditative or mind-body intervention (e.g., mindfulness, yoga)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) Pain Interference subscale | Change from baseline to 3-month follow-up
  Self-report questionnaire; pain interference subscale includes 7 items measuring the degree to which pain interferes with various aspects of life, including mobility, social activities, and mood. Subscale scores range from 0 to 70 with higher scores indicative of greater pain disability.
Clinical Global Impression scale (CGI) | Change from baseline to 3-month follow-up
  The CGI consists of two clinician-rated one-item measures assessing 1) the severity of psychopathology from 1 (normal, not at all ill) to 7 (among the most extremely ill patients), CGI-S, and 2) the improvement in functioning since baseline assessment from 1 (very much improved since the initiation of treatment) to 7 (very much worse since the initiation of treatment), CGI-I. The CGI is a well-established measure of psychological symptom severity and is applicable across psychological conditions.

SECONDARY OUTCOMES:
Satisfaction with Life Scale (SWLS) | Change from baseline to 3-month follow-up
  Self-report questionnaire; 5 items assessing global life satisfaction. Total scores range from 5 to 35, with higher scores indicating greater satisfaction with life.
Veterans SF-36 | Change from baseline to 3-month follow-up
  Self-report questionnaire with 36 items that assesses health-related quality of life; yields a physical component summary (PCS) and a mental component summary (MCS).

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Malaktaris, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Specific parameters of sharing are not yet established

DOCUMENTS (1):
  • Informed Consent Form (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT04651296/ICF_000.pdf